CLINICAL TRIAL: NCT03882944
Title: A Prospective, Observational Study of the Effect of a High Calorie and Protein Oral Nutritional Supplement, in an Older Malnourished or at Risk of Malnutrition, Hip Fracture Population
Brief Title: An Observational Study of a Nutritional Supplement in an Older Malnourished or at Risk of Malnutrition, Hip Fracture Population
Status: Completed | Type: Observational
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Other Study IDs: DA20
Record Dates: First submitted 2019-03-06; First posted 2019-03-20 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This non-interventional, prospective, observational study is designed to observe the use of high calorie, high protein oral nutritional supplement in malnourished or at risk of malnutrition patients after hip fracture surgery, as assessed by a clinician. Subjects will be enrolled and observed for a period of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject has voluntarily signed and dated an informed consent form, approved by an Independent Ethics Committee, prior to any participation in the study.
* Subject is considered malnourished, or is at risk for malnutrition
* Subject conforms to the requirements set forth on the study product label.
* Subject has an estimated, or measured, glomerular filtration rate >30ml/min/1.73m2 (MDRD equation).
* Subject has been elected for hip fracture surgery and is within three days since surgery.
* The study physician determines the subject is fit to participate.
* Subject is under the care of a health care professional for malnutrition, or is at risk for malnutrition, and has recently been prescribed study oral nutritional supplement by their health care professional.
* After surgery, the subject is free living, resides in a nursing home, or remains in hospital and has an expected length of hospital stay < 15 days.

Exclusion Criteria:

* Subject has known dementia, brain metastases, eating disorders, history of significant neurological or psychiatric disorder, or any other psychological condition that may interfere with study product consumption AND does not have a caregiver who can assist them with adherence to the study protocol.
* Subject has active cancer and the study physician determines the subject is not suitable for the study.
* Subject has uncontrolled diabetes.
* Subject is known to be allergic or intolerant to any ingredient found in the study product.
* Participation in another study that has not been approved as a concomitant study.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population will include older men and women who are free living (outpatient) or residing in a nursing home, who meet all enrollment criteria. Subjects will be recruited by the investigator(s) from each study site.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
Nutritional Status | Baseline to Week 12
  Measured by the Mini Nutritional Assessment (MNA) 18 questions; 30 total point scale where lower number indicates risk of malnutrition

SECONDARY OUTCOMES:
Barthel Index of Activities of Daily Living | Baseline to Week 12
  Subject completed assessment of 10 functions; Sum of scores range from 0-100 scaled in positive direction
Functional Ambulation Classification Scale (FAC) | Baseline to Week 12
  6-level scale assesses ambulation status; scaled in the positive direction; the higher level indicates greater ambulation
Short Physical Performance Battery (SPPB) | Week 12
  Timed assessments of balance, gait speed and chair standing; Scaled in the negative direction
Compliance with Nutritional Supplement | Baseline to Week 12
  Subject completed consumption dairy

OTHER OUTCOMES:
Blood Chemistries - Chemistry Profile | Baseline to Week 12
  Blood chemistries collected per standard of care
Blood Chemistries - Hematology Profile | Baseline to Week 12
  Hematology blood chemistries collected per standard of care
Blood Chemistries - Lipid Panel | Baseline to Week 12
  Lipid panel blood chemistries collected per standard of care
Body Mass Index | Baseline to Week 12
  BMI calculated Weight (kg)/Height (m)2
Length of Stay in Hospital | Week 12
  Information collected for hospital admission and discharge dates
Healthcare provider satisfaction questionnaire | Week 12
  HCP completed questionnaire; 3 to 5 category responses scaled in negative direction
Subject satisfaction questionnaire | Week 12
  Subject completed questionnaire; Responses 1 to 10 scaled in the positive direction
Medication Use | Baseline to Week 12
  Medications prescribed

CONTACTS AND LOCATIONS:
Overall Officials: Maria Camprubi, PhD, Study Chair — Abbott
Locations (17):
- Spain (17):
  - Hospital de Alcorcón, Alcorcón
  - Complejo Asistencial de Avila, Ávila
  - Hospital Cruz Roja Gijón, Gijón
  - Hospital Universitario de Guadalajara, Guadalajara
  - Hospital Infanta Elena, Huelva
  - Hospital Universitario de Gran Canaria Doctor Negrin, Las Palmas
  - Complejo Asistencial Universitario de León, León
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Virgen del Puerto, Plasencia
  - Hospital Universitario De Salamanca, Salamanca
  - Hospital Nuestra Señora de Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario Dr. Peset, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid